CLINICAL TRIAL: NCT00208676
Title: Non-Invasive Quantitation of Myocardial Dysfunction by Tissue Doppler / Synchronization Imaging in Children With Congenital Heart Defects (CHD)
Brief Title: Using Tissue Doppler/Synchronization to Determine Heart Function in Children With Congenital Heart Disease
Status: Terminated | Type: Observational
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, William T. Mahle, MD, Principal Investigator, Emory University
Other Study IDs: 0807-2004
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2013-11-27 (Estimated); Status verified 2013-11

CONDITIONS: Congenital Heart Defects
Keywords: heart defects; pediatrics
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
There are many children that have heart dysfunction because they are either born with Congenital Heart Disease (CHD) or developed poor heart function because their hearts are ill. The invention of medical technology helps in the treatment of these children. New heart echocardiogram (echo) techniques including Tissue Doppler (TDI), Tissue Synchronization Imaging (TSI) and 3 dimensional echocardiography (3D) are imaging technologies that we hope will help in the diagnosis and treatment of these children.

Tissue Doppler Imaging is a noninvasive technique that measures the speed of heart muscle movement. Tissue Synchronization Imaging measures how well the lower pumping chambers of the heart are working together. A 3D echo is a 3 dimensional picture of a beating heart that allows your doctor to see the heart from any angle. These techniques are noninvasive, meaning on the outside of your body. The size and function of the ventricles (the lower part of the heart) can change under different conditions. Using these techniques we will attempt to better determine how well the ventricles function during illness and health.

DETAILED DESCRIPTION:
All subjects who are treated at Sibley Heart Center at Children's Healthcare of Atlanta with the diagnosis of a congenital heart defect or an acquired heart condition (i.e. heart failure) may be approached for possible participation into the study. These patients will include newly diagnosed patients as well as patients who were diagnosed in previous years and have received medical treatment for their defect or condition. The following describe study procedures:

Echocardiographic assessment Standard 2-dimensional, M-mode, and Doppler or 3-dimensional echocardiography evaluation will be performed. We will assess cardiac function using left ventricular shortening (SF) and ejection fractions (EF). The EF will be calculated using both M-Mode and by Simpson's rule. We will also perform tissue synchronization imaging (TSI) and tissue Doppler imaging (TDI) using the GE Vivid 7 echocardiographic system. Both TSI and TDI will assist investigators in assessing mechanical synchrony. The research echocardiograms will occur at the time of routine assessments.

Clinical assessment/data collection Clinical information from the chart will be collected for this study. The information will include the doctor's evaluation of general health, including diagnosis and the names of any medications the participant may be taking. If the child has undergone a routine MRI for the purpose of clinical care, the MRI measures will be collected in order to compare MRI images and measures to the new 3D echo technique. Finally, EKG data will be collected at each visit. EKGs are performed routinely for these patients however, if one is not performed, the study staff will perform an EKG assessment in order to have electromechanical information (i.e. arrhythmias) on all children participating.

ELIGIBILITY:
Inclusion Criteria:

Any child up to 21 years of age with a congenital heart defect -

Exclusion Criteria:

-

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 200
Dates: Start 2005-09; Study Completion 2006-01

CONTACTS AND LOCATIONS:
Overall Officials: Derek Fyfe, MD, Principal Investigator — Emory University
Locations (1):
- Children's Healthcare of Atlanta at Egleston, Atlanta, Georgia, United States

REFERENCES:
- [Background] Hibberd MG, Chuang ML, Beaudin RA, Riley MF, Mooney MG, Fearnside JT, Manning WJ, Douglas PS. Accuracy of three-dimensional echocardiography with unrestricted selection of imaging planes for measurement of left ventricular volumes and ejection fraction. Am Heart J. 2000 Sep;140(3):469-75. doi: 10.1067/mhj.2000.108513. PMID 10966550
- [Background] Chuang ML, Parker RA, Riley MF, Reilly MA, Johnson RB, Korley VJ, Lerner AB, Douglas PS. Three-dimensional echocardiography improves accuracy and compensates for sonographer inexperience in assessment of left ventricular ejection fraction. J Am Soc Echocardiogr. 1999 May;12(5):290-9. doi: 10.1016/s0894-7317(99)70049-0. PMID 10231614